CLINICAL TRIAL: NCT03143166
Title: Relative Bioavailability of Tablet Formulation of Dabigatran Etexilate With and Without Co-administration of Rabeprazole in Healthy Male Subjects (an Open-label, Single-dose, Two-period, Single-arm Study)
Brief Title: Pradaxa Tablet Proton Pump Inhibitor (PPI) Bioavailability (BA) Study in Japan
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1160-0270
Record Dates: First submitted 2017-05-04; First posted 2017-05-08 (Actual); Results first posted 2019-01-16 (Actual); Last update posted 2019-01-16 (Actual); Status verified 2018-07

CONDITIONS: Non-alcoholic Fatty Liver Disease
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease | interventions — Dabigatran; Telmisartan

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- All participants (Experimental): Dabigatran etexilate given without rabeprazole and then Dabigatran etexilate given without rabeprazole.
  Interventions: Drug: Dabigatran Etexilate; Drug: Rabeprazol sodium

INTERVENTIONS:
Drug: Dabigatran Etexilate — Tablet, film coated
  Other Names: MICARDIS, PRITOR, TELMISARTAN
Drug: Rabeprazol sodium — Tablet

SUMMARY:
The primary objective of this trial is to investigate the relative Bioavailability (BA) of tablet formulation of Dabigatran etexilate (DE) with and without co-administration of rabeprazole in healthy male subjects.

The secondary objective is the evaluation and comparison of several pharmacokinetic parameters between the treatments.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male subjects according to the investigator's assessment, based on a complete medical history including a physical examination, vital signs (blood pressure (BP), pulse rate (PR)), 12-lead electrocardiogram (ECG), and clinical laboratory tests
* Age ≥ 20 and ≤ 40 years at informed consent
* Body mass index (BMI) of 18 ≥ and ≤ 25 kg/m2 at screening
* Signed and dated written informed consent prior to admission to the study in accordance with Good Clinical Practice (GCP) and local legislation

Exclusion Criteria:

* Any finding in the medical examination (including blood pressure (BP), pulse rate (PR) or electrocardiogram (ECG)) is deviating from normal and judged as clinically relevant by the investigator
* Measurement of systolic blood pressure (BP) outside the range of 90 to 140 mmHg, diastolic blood pressure outside the range of 50 to 90 mmHg, or pulse rate (PR) outside the range of 45 to 90 bpm at screening
* Any laboratory value outside the reference range before administration of DE that the investigator considers to be of clinical relevance
* Any evidence of a concomitant disease judged as clinically relevant by the investigator
* Any relevant bleeding history considered by the investigator
* Any history or evidence of blood dyscrasia, haemorrhagic diathesis, severe thrombocytopenia, cerebrovascular haemorrhage, bleeding tendencies associated with active ulceration or overt bleeding of gastrointestinal, respiratory or genitourinary tract or any disease or condition with haemorrhagic tendencies
* Gastrointestinal, hepatic, renal, respiratory, cardiovascular, metabolic, immunological or hormonal disorders
* Any history of hypochlorhydria or achlorhydria
* Cholecystectomy and/or surgery of the gastrointestinal tract that could interfere with the pharmacokinetics of the trial medication (except appendectomy and simple hernia repair)
* Planned surgeries within four weeks following the end-of trial examination
* Diseases of the central nervous system (including but not limited to any kind of seizures or stroke), and other relevant neurological or psychiatric disorders
* History of relevant orthostatic hypotension, fainting spells, or blackouts
* Chronic or relevant acute infections
* History of relevant allergy or hypersensitivity (including allergy to the trial medication or its excipients)
* Use of drugs within 30 days prior to administration of trial medication if that might reasonably influence the results of the trial (incl. QT/QTc interval prolongation)
* Participation in another trial where an investigational drug has been administered within 60 days prior to planned administration of trial medication, or current participation in another trial involving administration of investigational drug
* Smoker (more than 10 cigarettes or 3 cigars or 3 pipes per day)
* Inability to refrain from smoking at trial site
* Alcohol abuse (consumption of more than 30 g per day: e.g., 750 ml of beer, 1.5 gous [equivalent to 270 mL] of Sake)
* Drug abuse or positive drug screening
* Blood donation of more than 100 mL within 30 days prior to administration of trial medication or intended donation during the trial
* Intention to perform excessive physical activities within one week prior to administration of trial medication or during the trial
* Inability to comply with dietary regimen of trial site
* Subject is assessed as unsuitable for inclusion by the investigator, for instance, because considered not able to understand and comply with study requirements, or has a condition that would not allow safe participation in the study

Ages: 20 Years to 40 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2017-05-22 (Actual); Primary Completion 2017-07-27 (Actual); Study Completion 2017-08-02 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Souseikai Hakata Clinic, Fukuoka, Fukuoka, Japan

REFERENCES:
- [Derived] Harada A, Ikushima I, Haranaka M, Yanagihara A, Nakayama D. Bioequivalence of a Newly Developed Dabigatran Etexilate Tablet Versus the Commercial Capsule and Impact of Rabeprazole-Induced Elevated Gastric pH on Exposure in Healthy Subjects. Am J Cardiovasc Drugs. 2020 Jun;20(3):249-258. doi: 10.1007/s40256-019-00377-x. PMID 31667735

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This was open label, 2 period, fixed sequence (RT), single arm study in 36 healthy male Japanese subjects. All subjects were orally treated with single dose of 110 milligram (mg) dabigatran etexilate (DE) tablet formulation alone in period 1 and with 20 mg rabeprazole tablet in period 2 with 4 days of rabeprazole pre-medication.
Pre-assignment Details: After it had been determined that the subject met all eligibility criteria, a unique subject number was assigned. The number was recorded on electronic Case Report Forms and correspondence regarding the subject. Once a subject number had been assigned, it could not be reassigned to any other subject. Randomisation was not planned in this study.
Groups:
- Dabigatran Etexilate 110 mg With and Without Rabeprazole 20 mg: Subjects were treated orally with dabigatran etexilate 110 mg tablet alone (Reference) after an overnight fast of at least 10 hours (h) without pretreatment with rabeprazole 20 mg tablet in period 1 followed by single dose of dabigatran etexilate 110 mg tablet and rabeprazole 20 mg tablets (Test) once daily with 4 days of rabeprazole pre-treatment in period 2. The treatments of dabigatran etexilate were separated by a wash-out phase of at least 4 days.
Period: Period 1
Arm/Group | Dabigatran Etexilate 110 mg With and Without Rabeprazole 20 mg
Started | 36
Completed | 36
Not Completed | 0
Period: Period 2 (Washout of at Least 4 Days)
Arm/Group | Dabigatran Etexilate 110 mg With and Without Rabeprazole 20 mg
Started | 36
Completed | 35
Not Completed | 1
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Population: Treated set (TS) : All enrolled subjects provided with trial medication and documented to have taken at least 1 dose of trial medication were included in the TS.
Groups:
- Total Subjects: Subjects were treated orally with dabigatran etexilate 110 mg tablet alone (Reference) after an overnight fast of at least 10 hours (h) without pretreatment with rabeprazole 20 mg tablet in period 1 followed by single dose of dabigatran etexilate 110 mg tablet and rabeprazole 20 mg tablets (Test) once daily with 4 days of rabeprazole pre-treatment in period 2. The treatments of dabigatran etexilate were separated by a wash-out phase of at least 4 days.
Arm/Group | Total Subjects
Number analyzed (Participants) | 36
Age, Continuous [Mean (Standard Deviation); unit: Years] — Age of all subjects enrolled in the study. Population: TS
  Years | 26.3 (4.7)
Sex: Female, Male [Count of Participants; unit: Participants] — Gender distribution of all subjects enrolled in the study. Population: TS
  Participants
    Female | 0
    Male | 36
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Ethnicity of all subjects enrolled in the study. Population: TS
  Participants
    Hispanic or Latino | 0
    Not Hispanic or Latino | 36
    Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants] — Race of all subjects enrolled in the study. Population: TS
  Participants
    American Indian or Alaska Native | 0
    Asian | 36
    Native Hawaiian or Other Pacific Islander | 0
    Black or African American | 0
    White | 0
    More than one race | 0
    Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Area Under the Plasma Concentration-time Curve From 0 to Time of Last Quantifiable Time Point (tz) of Total Dabigatran (AUC0-tz).
Description: This endpoint calculates area under the concentration-time curve of total dabigatran in plasma over the time interval from 0 to the time of last quantifiable time point.
Time Frame: Samples were collected 1 hour Pre-dose and at 0:30, 1:00, 1:30, 2:00, 3:00, 4:00, 6:00, 8:00, 12:00, 24:00 36:00 and 48:00 hours post dose.
Population: Pharmacokinetic set (PKS): All treated subjects who provided at least 1 observation for at least 1 primary endpoint without important protocol violations with respect to the statistical evaluation of Pharmacokinetic (PK) endpoints were included in PKS.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Nanogram*Hour/ millilitre (ng*h/mL)
Groups:
- Dabigatran Etexilate 110 mg (Reference): Subjects were treated orally with dabigatran etexilate 110 mg tablet alone after an overnight fast of at least 10 hours (h) without pre-treatment with rabeprazole 20 mg tablet.
- Dabigatran Etexilate 110 mg + Rabeprazole 20 mg Tablet (Test): Subjects were treated orally with single dose of dabigatran etexilate 110 mg tablet and rabeprazole 20 mg tablets once daily with 4 days of rabeprazole pre-treatment.
Arm/Group | Dabigatran Etexilate 110 mg (Reference) | Dabigatran Etexilate 110 mg + Rabeprazole 20 mg Tablet (Test)
Number analyzed (Participants) | 36 | 35
Nanogram*Hour/ millilitre (ng*h/mL) | 667 (123) | 192 (109)
Statistical Analysis 1: Comparison: Dabigatran Etexilate 110 mg (Reference) vs Dabigatran Etexilate 110 mg + Rabeprazole 20 mg Tablet (Test); Test type: Other; ANOVA; An analysis of variance (ANOVA) was used on the logarithmic scale including effects for 'subjects' and 'treatment'; Adjusted gMean ratio Test/Reference (%) = 28.85, 90% CI 2-sided [21.346 to 38.996], Standard Error of Mean 86.7 — The dispersion value standard error of the mean is actually intra individual geometric coefficient of variation (gCV) (%)

2. Primary Outcome: Maximum Concentration of Total Dabigatran in Plasma (Cmax).
Description: This outcome is maximum measured concentration of the total dabigatran in plasma
Time Frame: as for outcome 1
Population: PKS
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Nano gram per milliliter (ng/mL)
Arm/Group | Dabigatran Etexilate 110 mg (Reference) | Dabigatran Etexilate 110 mg + Rabeprazole 20 mg Tablet (Test)
Number analyzed (Participants) | 36 | 35
Nano gram per milliliter (ng/mL) | 83.1 (118) | 21.8 (105)
Statistical Analysis 1: Comparison: Dabigatran Etexilate 110 mg (Reference) vs Dabigatran Etexilate 110 mg + Rabeprazole 20 mg Tablet (Test); Test type: Other; ANOVA; An analysis of variance (ANOVA) was used on the logarithmic scale including effects for 'subjects' and 'treatment'; Adjusted gMean ratio Test/Reference (%) = 26.37, 90% CI 2-sided [20.066 to 34.665], Standard Error of Mean 76.6 — [estimate comment as in outcome 1, analysis 1]

3. Secondary Outcome: Area Under the Plasma Concentration-time Curve From 0 to Time of Last Quantifiable Time Point (tz) of Free Dabigatran (AUC0-tz).
Description: This endpoint calculates area under the concentration-time curve of free dabigatran in plasma over the time interval from 0 to the time of last quantifiable time point.
Time Frame: as for outcome 1
Population: PKS
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Nanogram*Hour/ millilitre (ng*h/mL)
Arm/Group | Dabigatran Etexilate 110 mg (Reference) | Dabigatran Etexilate 110 mg + Rabeprazole 20 mg Tablet (Test)
Number analyzed (Participants) | 36 | 35
Nanogram*Hour/ millilitre (ng*h/mL) | 588 (119) | 164 (110)
Statistical Analysis 1: Comparison: Dabigatran Etexilate 110 mg (Reference) vs Dabigatran Etexilate 110 mg + Rabeprazole 20 mg Tablet (Test); Test type: Other; ANOVA; An analysis of variance (ANOVA) was used on the logarithmic scale including effects for 'subjects' and 'treatment'; Adjusted gMean ratio Test/Reference (%) = 28.02, 90% CI 2-sided [20.914 to 37.537], Standard Error of Mean 83.4 — [estimate comment as in outcome 1, analysis 1]

4. Secondary Outcome: Maximum Concentration of Free Dabigatran in Plasma (Cmax).
Description: This outcome is maximum measured concentration of the free dabigatran in plasma
Time Frame: as for outcome 1
Population: PKS
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Nanogram per milliliter (ng/mL)
Arm/Group | Dabigatran Etexilate 110 mg (Reference) | Dabigatran Etexilate 110 mg + Rabeprazole 20 mg Tablet (Test)
Number analyzed (Participants) | 36 | 35
Nanogram per milliliter (ng/mL) | 72.9 (114) | 20.0 (103)
Statistical Analysis 1: Comparison: Dabigatran Etexilate 110 mg (Reference) vs Dabigatran Etexilate 110 mg + Rabeprazole 20 mg Tablet (Test); Test type: Other; ANOVA; An analysis of variance (ANOVA) was used on the logarithmic scale including effects for 'subjects' and 'treatment'; Adjusted gMean ratio Test/Reference (%) = 27.56, 90% CI 2-sided [21.023 to 36.118], Standard Error of Mean 75.6 — [estimate comment as in outcome 1, analysis 1]

5. Secondary Outcome: Area Under the Concentration-time Curve of Total Dabigatran in Plasma Over the Time Interval From 0 Extrapolated to Infinity (AUC0-∞).
Description: This endpoint calculates area under the concentration-time curve of total dabigatran in plasma over the time interval from 0 extrapolated to infinity
Time Frame: as for outcome 1
Population: PKS
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Nanogram*Hour/ millilitre (ng*h/mL)
Arm/Group | Dabigatran Etexilate 110 mg (Reference) | Dabigatran Etexilate 110 mg + Rabeprazole 20 mg Tablet (Test)
Number analyzed (Participants) | 36 | 35
Nanogram*Hour/ millilitre (ng*h/mL) | 702 (110) | 214 (96.6)
Statistical Analysis 1: Comparison: Dabigatran Etexilate 110 mg (Reference) vs Dabigatran Etexilate 110 mg + Rabeprazole 20 mg Tablet (Test); Test type: Other; ANOVA; An analysis of variance (ANOVA) was used on the logarithmic scale including effects for 'subjects' and 'treatment'; Adjusted gMean ratio Test/Reference (%) = 30.59, 90% CI 2-sided [23.260 to 40.234], Standard Error of Mean 76.8 — [estimate comment as in outcome 1, analysis 1]

6. Secondary Outcome: Area Under the Concentration-time Curve of Free Dabigatran in Plasma Over the Time Interval From 0 Extrapolated to Infinity (AUC0-∞).
Description: This endpoint calculates area under the concentration-time curve of free dabigatran in plasma over the time interval from 0 extrapolated to infinity.
Time Frame: as for outcome 1
Population: PKS
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Nanogram*Hour/ millilitre (ng*h/mL)
Arm/Group | Dabigatran Etexilate 110 mg (Reference) | Dabigatran Etexilate 110 mg + Rabeprazole 20 mg Tablet (Test)
Number analyzed (Participants) | 36 | 35
Nanogram*Hour/ millilitre (ng*h/mL) | 618 (107) | 188 (93.4)
Statistical Analysis 1: Comparison: Dabigatran Etexilate 110 mg (Reference) vs Dabigatran Etexilate 110 mg + Rabeprazole 20 mg Tablet (Test); Test type: Other; ANOVA; An analysis of variance (ANOVA) was used on the logarithmic scale including effects for 'subjects' and 'treatment'; Adjusted gMean ratio Test/Reference (%) = 30.61, 90% CI 2-sided [23.404 to 40.037], Standard Error of Mean 74.9 — [estimate comment as in outcome 1, analysis 1]

ADVERSE EVENTS:
Time Frame: From first drug administration until 3 days after the last drug administration. Up to 10 days.
Description: An adverse event (AE) was defined as any untoward medical occurrence in a subject or clinical investigation subject administered a medicinal product and which did not necessarily have to have a causal relationship with this treatment. Treated Set was used for assessment of AEs.
Groups:
- Dabigatran Etexilate 110 mg + Rabeprazole 20 mg (Test): Subjects were treated orally with single dose of dabigatran etexilate 110 mg tablet and rabeprazole 20 mg tablets once daily with 4 days of rabeprazole pre-treatment.
Arm/Group | Dabigatran Etexilate 110 mg (Reference) | Dabigatran Etexilate 110 mg + Rabeprazole 20 mg (Test)
All-Cause Mortality (participants affected / at risk) | 0/36 | 0/35
Serious Adverse Events (participants affected / at risk) | 0/36 | 0/35
Other Adverse Events (participants affected / at risk) | 0/36 | 0/35

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Boehringer Ingelheim (BI) acknowledges that investigators have the right to publish the study results. Investigators shall provide BI with a copy of any publication or presentation for review prior to any submission. Such review will be done with regard to proprietary information, information related to patentable inventions, medical, scientific, and statistical accuracy within 60 days. BI may request a delay of the publication in order to protect BI's intellectual property rights.

DOCUMENTS (2):
  • Statistical Analysis Plan (2017-08-23): https://cdn.clinicaltrials.gov/large-docs/66/NCT03143166/SAP_000.pdf
  • Study Protocol (2017-04-20): https://cdn.clinicaltrials.gov/large-docs/66/NCT03143166/Prot_001.pdf